CLINICAL TRIAL: NCT01207037
Title: Study of Prognostic Factors of Acute Splenic Sequestration in a Cohort of Sickle Cell Disease (SCD) Children Diagnosed at Birth
Brief Title: Prognostic Factors of Acute Splenic Sequestration
Acronym: SSADREPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P071228; 2009-A00142-55 (Other: AFSSAPS)
Record Dates: First submitted 2010-06-03; First posted 2010-09-22 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Anemia; Drepanocytic
MeSH Terms: conditions — Anemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other)
  Interventions: Procedure: blood samples and scintigraphy

INTERVENTIONS:
Procedure: blood samples and scintigraphy — at 3 months, 6 months, 12 months, 18 months and 24 months will allow a clinical evaluation and an additional sampling of blood of 5 mL at each visit Scintigraphy at 6 months and 18 months

SUMMARY:
Acute splenic sequestration is a frequent and life threatening complication occurring in approximately 10 % of homozygous children. Maximal incidence is between 6 and 18 months.

The investigators formulate the hypothesis that there are clinical, biological and genetic markers predictive of severe complications notably acute splenic sequestration in SCD children. The present research project thus aims at analyzing in a forward-looking way the profile of severity by analysing clinical, biological and genetic characteristics in a multicentric cohort of 60 SCD children

DETAILED DESCRIPTION:
A prospective multicentric analysis will be conducted in a cohort of 150 SS or S ß ° children diagnosed at birth, included at 3 -5 months and followed up to the age of 24 months.

Five visits, superimposed to the usual follow-up of SCD children, (Recommendations of the High Authority of Health) at 3 months, 6 months, 12 months, 18 months and 24 months will allow a clinical evaluation and an additional sampling of blood (5 mL) at each visit.

The samples will allow 1.analysis of the red blood cell phenotype (adhesion and deformability) and densities 2. the genetic profile 3.to establish a cell bank, a sera bank and a DNA bank, Spleen function in the cohort will be estimated by spleen scintigraphy, coupled with blood markers (pitted cells, Howell-Jolly bodies counts)

ELIGIBILITY:
Inclusion criteria :

* Children aged 3 to 6 months
* homozygous (SS) or S beta° sickle cell disease diagnosed by neonatal screening
* With no history of acute splenic sequestration
* Signed parental consent
* Patient covered by national insurance scheme or CMU

Exclusion criteria :

* Children with other SCD genotype
* Children with congenital anatomical asplenia
* Children with previous episode of acute splenic sequestration
* Absence of possible follow-up
* Simultaneous enrolment in another biomedical research

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2010-08-12 (Actual); Primary Completion 2014-12-22 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Study of prognostic factors of acute splenic sequestration | after three years
  * Complete blood count, reticulocyte count, haemoglobin level, VGM, TGMH, CCMH, hematocrit, % foetal haemoglobin (HbF), red blood cell densities (2 mL)
  * Deformability of red blood cells
  * Expression study of the cell surface molecule: Phosphatidyl serine, CD 36, READ B-CAM, CD 47, ICAM 4, VLA 4. (Cellulotheque = red blood cells frozen in cryopreservative conditions)
  * Total LDH, Bilirubine (stigmas of hemolysis)
  * Genetic Profil ( DNAtheque)

SECONDARY OUTCOMES:
Study of hematology parameters | after three years
  * Percentage of Howell Jolly's bodies (0,1 mL)
  * Percentage of pitted cells (0,5 mL fixed in 4 %)formaldehyde
  * Splenic volume, semi-quantitative measure in scintigraphy
  * Antibody titers in answer to the antipneumococcic vaccination ( serotheque)

CONTACTS AND LOCATIONS:
Overall Officials: Valentine Brousse, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Necker Hospital, Paris, France

REFERENCES:
- [Background] El Hoss S, Cochet S, Marin M, Lapoumeroulie C, Dussiot M, Bouazza N, Elie C, de Montalembert M, Arnaud C, Guitton C, Pellegrino B, Odievre MH, Moati F, Le Van Kim C, Aronovicz YC, El Nemer W, Brousse V. Insights into determinants of spleen injury in sickle cell anemia. Blood Adv. 2019 Aug 13;3(15):2328-2336. doi: 10.1182/bloodadvances.2019000106. PMID 31391165
- [Background] Brousse V, El Hoss S, Bouazza N, Arnaud C, Bernaudin F, Pellegrino B, Guitton C, Odievre-Montanie MH, Mames D, Brouzes C, Picard V, Nguyen-Khoa T, Pereira C, Lapoumeroulie C, Pissard S, Gardner K, Menzel S, Le Van Kim C, Colin-Aronovicz Y, Buffet P, Mohandas N, Elie C, Maier-Redelsperger M, El Nemer W, de Montalembert M. Prognostic factors of disease severity in infants with sickle cell anemia: A comprehensive longitudinal cohort study. Am J Hematol. 2018 Nov;93(11):1411-1419. doi: 10.1002/ajh.25260. Epub 2018 Sep 21. PMID 30132969
- [Background] Brousse V, Colin Y, Pereira C, Arnaud C, Odievre MH, Boutemy A, Guitton C, de Montalembert M, Lapoumeroulie C, Picot J, Le Van Kim C, El Nemer W. Erythroid Adhesion Molecules in Sickle Cell Anaemia Infants: Insights Into Early Pathophysiology. EBioMedicine. 2014 Dec 18;2(2):154-7. doi: 10.1016/j.ebiom.2014.12.006. eCollection 2015. PMID 26137540